CLINICAL TRIAL: NCT06557096
Title: Open-label, Single-Arm, Multicenter Clinical Study of EGFR-TKIs Sequentially Combined With Bevacizumab for the Treatment of EGFR-Mutant Advanced Non-Small Cell Lung Cancer, Based on Early Warning by CSF CTC Capture Technology
Brief Title: CSF CTC-Capture-Guided EGFR-TKI and Bevacizumab Combination Therapy in EGFR-Mutant Advanced NSCLC
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2024-7604A
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-07

CONDITIONS: Non Small Cell Lung Cancer; Circulating Tumor Cell; EGF-R Positive Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplastic Cells, Circulating | interventions — osimertinib; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sequential Treatment cohort (Experimental): Participants receive osimertinib orally at a dose of 80mg daily for a 28-day treatment period. After the start of treatment, cerebrospinal fluid is collected every 12 weeks for circulating tumor cell (CTC) examination and routine cytopathological assessment. If the routine cytopathological test is positive, participants are sequentially treated with continued osimertinib at 80mg daily, in combination with bevacizumab administered intravenously at a dosage of 7.5mg/kg of body weight, on the first day of each cycle, with medication given once every 3 weeks. A continuous treatment of 21 days constitutes one treatment cycle. After the initiation of treatment, cerebrospinal fluid is collected every 6 weeks for CTC testing and routine cytopathological examination.
  Interventions: Drug: Osimertinib 80 MG; Drug: Bevacizumab

INTERVENTIONS:
Drug: Osimertinib 80 MG — Osimertinib is taken orally at a dose of 80mg daily for a 28-day treatment period, followed by a sequential treatment of osimertinib 80mg daily taken orally for another 28 days.
  Other Names: Tagrisso
Drug: Bevacizumab — Sequential combination therapy with bevacizumab administered intravenously at a dosage of 7.5mg/kg of body weight on the first day of each cycle, with medication given once every 3 weeks, for a continuous treatment duration of 21 days.
  Other Names: avastin

SUMMARY:
clinical trial The goal of this clinical trial is to learn whether the treatment of advanced non-small cell lung cancer with EGFR-TKIs, when combined with bevacizumab in the presence of positive circulating tumor cells in the cerebrospinal fluid, has better therapeutic efficacy. The main questions it aims to answer are:1.When EGFR-TKIs are sequentially combined with bevacizumab along with EGFR-TKIs for first-line treatment of advanced non-small cell lung cancer, how long can the participants survive? 2.What medical problems do participants have when using EGFR-TKIs sequentially combined with bevacizumab in conjunction with EGFR-TKIs.

Participants will:

Receive EGFR-TKIs treatment for a duration of 3 months, and upon a positive cerebrospinal fluid tumor cell status, subsequently receive bevacizumab combined with EGFR-TKIs treatment until disease progression.

Visit the clinic for check-ups and tests every two weeks, and have follow-up visits every six weeks after the treatment ends.

Keep a record of their symptoms and disease progression.

DETAILED DESCRIPTION:
This study is an open-label, single-arm, multicenter, exploratory clinical trial designed to evaluate and observe the first-line treatment of locally advanced/advanced non-small cell lung cancer that is positive for EGFR mutations, based on the early warning of a novel cerebrospinal fluid CTC capture technology. Subjects who meet all inclusion criteria and none of the exclusion criteria will first receive EGFR-TKIs (osimertinib, amivantamab, or futibatinib) treatment (as per the instruction manual). After a positive cerebrospinal fluid tumor cell status, they will then sequentially receive bevacizumab (7.5mg/kg, intravenous injection, once every 3 weeks) combined with EGFR-TKIs treatment.

Participants Aged 18 years or older (including 18 years old) and up to 75 years of age (including 75 years old); confirmed non-small cell lung cancer through histology or cytology; confirmed EGFR sensitive mutation (exon 19 deletion or L858R) prior to treatment; planned to receive first-line monotherapy with EGFR-TKIs (osimertinib, amivantamab, or futibatinib).

This study is an open-label, single-arm, multicenter, exploratory clinical trial. The primary research objective is to evaluate the overall survival time (OS) of patients with locally advanced/advanced EGFR-mutant non-small cell lung cancer (NSCLC) treated with EGFR tyrosine kinase inhibitors (EGFR-TKIs) sequentially combined with bevacizumab as a first-line treatment, based on the early warning of a novel cerebrospinal fluid circulating tumor cell (CSF CTC) capture technology. The study endpoint is the overall survival time (OS) of the patients. Referring to the results of our team's prospective study data and historical literature review study data, it is anticipated that the hazard ratio (HR) for overall survival (OS) of EGFR-TKIs sequentially combined with bevacizumab compared to EGFR-TKIs as a first-line treatment for high-risk patients with EGFR-mutant locally advanced/advanced NSCLC and leptomeningeal metastasis will be 0.78 (median OS improved from 18 months to 21 months). After the first subject is enrolled, with the longest observation period being 24 months, α set at two-sided 0.05, and a power of 80%, calculating with a 25% CSF tumor cell positivity rate and a 10% loss to follow-up rate, using the NCSS&PASS 15.0 software and the single-sample Logrank test method, after sample correction, this study plans to enroll approximately 100 subjects.

Based on the investigator-assessed Overall Survival (OS) as the primary efficacy endpoint, the median survival time will be estimated using the Kaplan-Meier method, and the median event time along with its two-sided 95% confidence interval will be presented. Additionally, the hazard ratio and its 95% confidence interval will be estimated as the main analysis.

ELIGIBILITY:
Inclusion Criteria:

* 1.The subjects voluntarily joined this study and signed the informed consent form, showing good compliance and cooperation with follow-up.

  2.Ages between 18 years old (inclusive) and 75 years old (inclusive). 3.ECOG score: 0-2 points. 4.Expected survival of no less than 3 months. 5.According to the RECIST 1.1 criteria, the patient has at least one extracranial target lesion.

  6.Diagnosed with non-small cell lung cancer based on histology or cytology. 7.No leptomeningeal metastasis (EANO criteria). 8.The tumor tissue samples or blood samples are confirmed to have EGFR-sensitive mutations (including exon 19 deletions or L858R).

  9.Have not received systemic anti-tumor treatment, and are planned to receive first-line monotherapy with osimertinib, aumolertinib, or furmonertinib.

  10.The main organ functions are normal, that is, they meet the following criteria:
  1. The standard for routine blood test should meet: HB≥90 g/L; ANC≥1.5×10^9/L; PLT≥80×10^9/L.
  2. The biochemical examination should meet the following standards: TBIL<1.5×ULN; ALT and AST<2.5×ULN; serum Cr≤1.25×ULN or endogenous creatinine clearance > 45 ml/min (Cockcroft-Gault formula). 11.Women of childbearing age must have taken reliable contraceptive measures and have undergone a pregnancy test (serum or urine) within 7 days before enrollment, with a negative result, and must be willing to use appropriate methods of contraception during the trial period and for 8 weeks after the last administration of the trial medication. For men, they must agree to use appropriate methods of contraception during the trial period and for 8 weeks after the last administration of the trial medication or have undergone surgical sterilization.

Exclusion Criteria:

1. Subjects have received any of the following treatments:

   1. Previously used any EGFR tyrosine kinase inhibitors;
   2. Previously received any chemotherapy for lung cancer;
   3. Previously received any radiotherapy for lung cancer (except for palliative radiotherapy for bone metastases);
   4. Within 4 weeks before the first administration of the study medication, the subject had undergone major surgery;
   5. Within 7 days before the first administration of the study medication, used strong inhibitors or inducers of CYP3A4.
2. Subjects with concurrent other malignant tumors, except for basal cell carcinoma of the skin and in situ cancer.
3. Subjects have uncontrollable malignant pleural effusion and pericardial effusion.
4. Subjects who are allergic to contrast agents used in CT and MRI or who cannot tolerate MRI examinations.
5. As judged by the investigator, there are any serious or poorly controlled systemic diseases, such as poorly controlled hypertension, active bleeding diathesis, or active infection.
6. Clinically severe gastrointestinal dysfunction that may affect the intake, transport, or absorption of medication, such as the inability to take oral medication, uncontrollable nausea or vomiting, a history of extensive gastrointestinal resection, untreated recurrent diarrhea, atrophic gastritis, gastric diseases requiring long-term use of proton pump inhibitors that have not been cured, Crohn's disease, ulcerative colitis, etc.
7. Hepatic encephalopathy, hepatorenal syndrome, or liver cirrhosis.
8. Meet any of the following cardiac examination results:

   1. The average value of the corrected QT interval (QTcF) derived from three electrocardiograms (ECG) at rest using the Fridericia formula is > 470 msec;
   2. Resting ECG indicates conduction or ECG morphological abnormalities (such as complete left bundle branch block, third-degree atrioventricular block, second-degree atrioventricular block, and PR interval > 250 msec, etc.);
   3. There are any factors that increase the risk of QTc prolongation or arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or any concomitant medication of unexplained sudden death in direct relatives under 40 years old or prolonged QT interval;
   4. The left ventricular ejection fraction (LVEF) is < 50%.
9. Insufficient bone marrow reserve or organ function, meeting any of the following laboratory limits:

   1. Absolute neutrophil count <1.5×10^9/L;
   2. Platelet count <100×10^9/L;
   3. Hemoglobin <90 g/L (<9 g/dL);
   4. If there is no clear liver metastasis, alanine aminotransferase (ALT) > 3 times the upper limit of normal (ULN); if there is liver metastasis, ALT > 5×ULN;
   5. If there is no clear liver metastasis, aspartate aminotransferase (AST) > 3×ULN; if there is liver metastasis, AST > 5×ULN;
   6. If there is no clear liver metastasis, total bilirubin > 1.5×ULN; or with Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastasis, total bilirubin > 3×ULN;
   7. Creatinine > 1.5×ULN and creatinine clearance <50 mL/min (calculated by the Cockcroft-Gault formula); creatinine clearance is only required to be confirmed if creatinine > 1.5×ULN;
   8. Serum albumin (ALB) <28 g/L.
10. Active fungal, bacterial, and/or viral infections requiring systemic treatment.
11. Female subjects who are pregnant, breastfeeding, or planning to become pregnant during the study period.
12. History of interstitial lung disease, drug-induced interstitial lung disease, history of radiation pneumonitis requiring steroid treatment, or any evidence of clinically active interstitial lung disease.
13. Subjects judged by the investigator to be likely non-compliant with the study procedures and requirements, such as those with a clear history of neurological or psychiatric disorders, or currently suffering from psychiatric disorders.
14. Subjects judged by the investigator to have any conditions that may endanger the subject's safety or interfere with the study assessment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival（OS） | From the start of therapy until death due to any cause, assessed up to 2 years after completion of treatment
  From the time of a patient's diagnosis or the commencement of treatment, to the time of the patient's death.Will be estimated using Kaplan-Meier product-limit method. The median OS times with two-sided 95% CIs will be estimated.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Within 8 weeks after completion of treatment
  Defined as the percentage of participants having an objective response (complete response [CR] or partial response [PR]), according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. The ORR of the drug will be assessed according to Simon's two stage design. The estimated ORR will be compared to the response rate specified in the null hypothesis (6%) using one-sided exact binomial test at type I error 5%. 95% confidence interval (C.I.) will be also reported.
Progression free survival (PFS) | From the start of therapy until disease progression, or death due to any cause, assessed up to 2 years after completion of treatment
  Will be determined by the immune complete response (iCR). Will be estimated using Kaplan-Meier product-limit method. The median PFS times with two-sided 95% CIs will be estimated.
Duration of Response (DOR) | Up to 2 years after completion of treatment
  Defined as the time from an initial objective response (CR or PR) according to RECIST v 1.1 until disease progression, or death due to any cause, as determined by iCR.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chuyang, Director, Study Director — Nanchang University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pisters KM, Le Chevalier T. Adjuvant chemotherapy in completely resected non-small-cell lung cancer. J Clin Oncol. 2005 May 10;23(14):3270-8. doi: 10.1200/JCO.2005.11.478. PMID 15886314
- [Background] Bonomi PD. Implications of key trials in advanced nonsmall cell lung cancer. Cancer. 2010 Mar 1;116(5):1155-64. doi: 10.1002/cncr.24815. PMID 20087963
- [Background] Gahr S, Stoehr R, Geissinger E, Ficker JH, Brueckl WM, Gschwendtner A, Gattenloehner S, Fuchs FS, Schulz C, Rieker RJ, Hartmann A, Ruemmele P, Dietmaier W. EGFR mutational status in a large series of Caucasian European NSCLC patients: data from daily practice. Br J Cancer. 2013 Oct 1;109(7):1821-8. doi: 10.1038/bjc.2013.511. Epub 2013 Sep 3. PMID 24002608
- [Background] Maemondo M, Inoue A, Kobayashi K, Sugawara S, Oizumi S, Isobe H, Gemma A, Harada M, Yoshizawa H, Kinoshita I, Fujita Y, Okinaga S, Hirano H, Yoshimori K, Harada T, Ogura T, Ando M, Miyazawa H, Tanaka T, Saijo Y, Hagiwara K, Morita S, Nukiwa T; North-East Japan Study Group. Gefitinib or chemotherapy for non-small-cell lung cancer with mutated EGFR. N Engl J Med. 2010 Jun 24;362(25):2380-8. doi: 10.1056/NEJMoa0909530. PMID 20573926
- [Background] Burtness B, Anadkat M, Basti S, Hughes M, Lacouture ME, McClure JS, Myskowski PL, Paul J, Perlis CS, Saltz L, Spencer S. NCCN Task Force Report: Management of dermatologic and other toxicities associated with EGFR inhibition in patients with cancer. J Natl Compr Canc Netw. 2009 May;7 Suppl 1:S5-21; quiz S22-4. doi: 10.6004/jnccn.2009.0074. PMID 19470276